CLINICAL TRIAL: NCT04429828
Title: PoWerS Study: Psychological Wellbeing for Healthcare Students: Evaluation of a COVID-19 Digital Learning Package
Brief Title: COVID-19 Psychological Wellbeing for Healthcare Students
Acronym: PoWerS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Holly Blake, Associate Professor of Behavioural Science, University of Nottingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PoWerS_June2020
Record Dates: First submitted 2020-06-11; First posted 2020-06-12 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Psychological Wellbeing
MeSH Terms: interventions — Health Personnel

STUDY DESIGN:
Intervention Model Description: All students have access to the COVID-19 educational package to support psychological wellbeing in healthcare students (usual practice). In this study the investigators will conduct semi-structured qualitative interviews with healthcare students about their mental wellbeing, and use of this e-package.
Masking Description: This is an evaluation of an educational learning package, which is a form of 'supportive intervention' for students provided during the coronavirus pandemic. Therefore the investigators will conduct interviews with people who have used the e-package. The investigators will interview up to 45 participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- e-package: psychological wellbeing for healthcare workers (Experimental): A COVID-19 educational package on psychological wellbeing for healthcare workers, accessible to all healthcare students.
  Interventions: Other: COVID-19 e-package: Psychological wellbeing for healthcare workers

INTERVENTIONS:
Other: COVID-19 e-package: Psychological wellbeing for healthcare workers — All healthcare students have access to a COVID-19 educational learning package around psychological wellbeing (usual practice). In this study the investigators will conduct semi-structured qualitative interviews with healthcare students about their mental wellbeing, and use of this e-package.

SUMMARY:
We have developed an online learning resource designed to support healthcare staff during and after the COVID-19 pandemic. This resource has been produced in anticipation of the psychological effect of working during this time. This is an open access, free, online resource available here: https://www.nottingham.ac.uk/toolkits/play_22794 It is designed to be relevant for healthcare staff, and we are evaluating it now with healthcare students as our next generation of healthcare staff. We are interested in knowing more about your views of healthcare students towards this package. This will help us to determine its value as a learning resource to support psychological wellbeing in healthcare students, alongside other welfare supports. The aim is to describe the views of healthcare students towards an e-learning package developed in response to COVID-19 on Psychological Wellbeing for Healthcare Workers.

DETAILED DESCRIPTION:
The investigators aim to:

* gather insight into the emotional highs and lows of being a healthcare student during the pandemic
* identify any facilitators, obstacles or barriers to accessing the e-package.
* identify perceptions of healthcare students towards the value of the e-package during and after the COVID19 pandemic.
* establish recommendations for longer-term support for psychological wellbeing in healthcare students.

Qualitative interviews will be conducted with up to 45 purposively sampled healthcare students who have accessed the e-learning resource. The interview will be semi-structured and include a measure of mental wellbeing (Warwick-Edinburgh Wellbeing Scale, 14-item - license received), and single items measures of job stressfulness, job satisfaction, presenteeism, turnover intentions and work engagement.

Findings will inform future supportive interventions for healthcare students.

ELIGIBILITY:
Inclusion criteria:

* Healthcare students (e.g. any students who are registered on a healthcare course).
* Ability to give informed consent.
* Ability to attend an individual interview (remotely).

Exclusion criteria:

• Not a registered healthcare student.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-06-13 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Qualitative Interviews with Healthcare Students | Once per study, telephone interview (during a 6-week interview period)
  Users of the e-package
Warwick-Edinburgh Mental Wellbeing Scale | Baseline
  14-item scale to measure mental wellbeing. Total scores range from 14 to 70 and higher scores indicate greater positive mental wellbeing.

SECONDARY OUTCOMES:
Single Item Measure of Global Job Stressfulness (Houdmont et al, 2019) | Baseline
  Single-item measure. Scores range from 1 to 5 and higher scores indicated greater job stressfulness.
Single Item Global Job Satisfaction Measure (Dolbier et al, 2005) | Baseline
  Single-item measure. Scores range from 1 to 5 and higher scores indicated greater job satisfaction.
Single Item Measure of Presenteeism (Aronsson & Gustafsson, 2004) | Baseline
  Single-item measure. Scores range from 1 to 4, with higher scores indicating greater presenteeism.
Single Item Measure of Turnover intentions | Baseline
  Single-item measure. Scored 1=no intent to leave, 2=intent to leave
Work Engagement (Shaufeli et al, 2006) | Baseline
  Dedication subscale of the 9-item Utrecht Work Engagement Scale (3 items will be used: 2, 3 and 4). Scores range from 0 to 6, with higher scores indicating greater work engagement.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Interview data will be made available on request (after study end).
Time Frame: Interview data will be available on request at study end (after publication of findings).
Access Criteria: On request.